CLINICAL TRIAL: NCT02656420
Title: Broccoli Sprout Dose Response: Bioavailability and Effects on Air Pollutants
Brief Title: Broccoli Sprout Dose Response: Bioavailability and Effects of Air Pollutants
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Qidong Liver Cancer Institute (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00006734; R01CA190610 (NIH)
Record Dates: First submitted 2016-01-05; First posted 2016-01-15 (Estimated); Results first posted 2019-05-01 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Environmental Carcinogenesis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebos (Placebo Comparator): Beverage (100 mL) containing pineapple juice, lime juice and water. Nightly for 10 days.
  Interventions: Drug: Placebos
- High Dose Broccoli Sprout (Experimental): Beverage (100 mL) containing glucoraphanin-rich (600 micromole) and sulforaphane-rich (40 micromole) broccoli sprout powder mixed in pineapple juice, lime juice and water. Nightly for 10 days.
  Interventions: Drug: Broccoli Sprout-derived Beverage
- Medium Dose Broccoli Sprout (Experimental): Beverage (100 mL) containing glucoraphanin-rich (300 micromole) and sulforaphane-rich (20 micromole) broccoli sprout powder mixed in pineapple juice, lime juice and water. Nightly for 10 days.
  Interventions: Drug: Broccoli Sprout-derived Beverage
- Low Dose Broccoli Sprout (Experimental): Beverage (100 mL) containing glucoraphanin-rich (120 micromole) and sulforaphane-rich (8 micromole) broccoli sprout powder mixed in pineapple juice, lime juice and water. Nightly for 10 days.
  Interventions: Drug: Broccoli Sprout-derived Beverage

INTERVENTIONS:
Drug: Broccoli Sprout-derived Beverage — Maximum, half and one-fifth doses of broccoli sprout-derived beverage compared to placebos.
  Arms: High Dose Broccoli Sprout; Low Dose Broccoli Sprout; Medium Dose Broccoli Sprout
Drug: Placebos — Placebo as comparison to broccoli sprout-derived beverages
  Arms: Placebos

SUMMARY:
This study will examine the extent to which lower doses of a broccoli-derived beverage enhance the detoxication of air pollutants excreted in urine as compared to an maximal dose shown to be effective previously.

DETAILED DESCRIPTION:
This is a 10-day placebo control Phase II broccoli sprout intervention to be conducted in Qidong, P.R. China. Up to twelve hundred people from the farming townships will be screened and one hundred seventy eligible individuals will be enrolled in the study. Participants will be randomized into 4 treatment groups: one will receive a juice beverage containing a standard dose of glucoraphanin- and sulforaphane-rich broccoli sprout powder mixed in pineapple juice, lime juice and water, the second will receive one-half dose, the third one-fifth dose and the fourth group will receive placebo beverage containing pineapple juice, lime juice and water. Participants will drink their assigned beverage every evening and provide consecutive 12-hour urine collections throughout the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* in good general health with no history of chronic illness
* normal liver function tests
* normal renal function tests

Exclusion Criteria:

* personal history of cancer except for non-melanoma skin cancer
* use of prescribed medicines
* for women, a positive pregnancy test

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2016-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kensler, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Qidong Liver Cancer Institute, Qidong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Egner PA, Chen JG, Zarth AT, Ng DK, Wang JB, Kensler KH, Jacobson LP, Munoz A, Johnson JL, Groopman JD, Fahey JW, Talalay P, Zhu J, Chen TY, Qian GS, Carmella SG, Hecht SS, Kensler TW. Rapid and sustainable detoxication of airborne pollutants by broccoli sprout beverage: results of a randomized clinical trial in China. Cancer Prev Res (Phila). 2014 Aug;7(8):813-823. doi: 10.1158/1940-6207.CAPR-14-0103. Epub 2014 Jun 9. PMID 24913818
- [Derived] Chen JG, Johnson J, Egner P, Ng D, Zhu J, Wang JB, Xue XF, Sun Y, Zhang YH, Lu LL, Chen YS, Wu Y, Zhu YR, Carmella S, Hecht S, Jacobson L, Munoz A, Kensler K, Rule A, Fahey J, Kensler T, Groopman J. Dose-dependent detoxication of the airborne pollutant benzene in a randomized trial of broccoli sprout beverage in Qidong, China. Am J Clin Nutr. 2019 Sep 1;110(3):675-684. doi: 10.1093/ajcn/nqz122. PMID 31268126

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Beverage (100 mL) containing pineapple juice, lime juice and water. Nightly for 10 days.
  Broccoli Sprout Powder: Maximum, half and one-fifth doses of broccoli sprout-derived beverage compared to placebo.
- High Dose Broccoli Sprout: Beverage (100 mL) containing glucoraphanin-rich (600 micromole) and sulforaphane-rich (40 micromole) broccoli sprout powder mixed in pineapple juice, lime juice and water. Nightly for 10 days.
  Broccoli Sprout Powder: Maximum, half and one-fifth doses of broccoli sprout-derived beverage compared to placebo.
- Medium Dose Broccoli Sprout: Beverage (100 mL) containing glucoraphanin-rich (300 micromole) and sulforaphane-rich (20 micromole) broccoli sprout powder mixed in pineapple juice, lime juice and water. Nightly for 10 days.
  Broccoli Sprout Powder: Maximum, half and one-fifth doses of broccoli sprout-derived beverage compared to placebo.
- Low Dose Broccoli Sprout: Beverage (100 mL) containing glucoraphanin-rich (120 micromole) and sulforaphane-rich (8 micromole) broccoli sprout powder mixed in pineapple juice, lime juice and water. Nightly for 10 days.
  Broccoli Sprout Powder: Maximum, half and one-fifth doses of broccoli sprout-derived beverage compared to placebo.
Period: Overall Study
Arm/Group | Placebo | High Dose Broccoli Sprout | Medium Dose Broccoli Sprout | Low Dose Broccoli Sprout
Started | 55 | 25 | 35 | 55
Completed | 55 | 24 | 35 | 55
Not Completed | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | High Dose Broccoli Sprout | Medium Dose Broccoli Sprout | Low Dose Broccoli Sprout | Total
Number analyzed (Participants) | 55 | 25 | 35 | 55 | 170
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 55 | 25 | 35 | 55 | 170
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 56 [53 to 61] | 59 [56 to 62] | 58 [50 to 64] | 60 [53 to 63] | 58 [50 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 18 | 28 | 43 | 127
  Male | 17 | 7 | 7 | 12 | 43
Region of Enrollment [Number; unit: participants]
  China | 55 | 25 | 35 | 55 | 170

OUTCOME MEASURES:

1. Primary Outcome: Sulforaphane Bioavailability Measured in Sequential 12-Hour Urine Samples
Description: Urinary excretion of broccoli-derived sulforaphane metabolites: sulforaphane-mercapturic acid. The metabolites were measured all 20 of the sequential 12-hour urine collections from each participant over the 10-day intervention period. Data from each individual were summed to provide a single "per 24-hours" value for each participant.
Time Frame: 10 days
Population: Placebo arm samples were not analyzed f because no sulforaphane was administered to this group. Historically, background levels from dietary sources in this population are very low compared to active intervention levels. In addition, one participant in the High Dose Broccoli Sprout arm did not complete the full protocol and was not included.
Measure: Geometric Mean (Inter-Quartile Range); unit: micromoles/24 hours
Arm/Group | Placebo | High Dose Broccoli Sprout | Medium Dose Broccoli Sprout | Low Dose Broccoli Sprout
Number analyzed (Participants) | 0 | 24 | 35 | 55
micromoles/24 hours |  | 24.8 [16.8 to 33.5] | 11.0 [8.4 to 13.2] | 4.3 [3.6 to 5.2]
Statistical Analysis 1: Comparison: High Dose Broccoli Sprout vs Medium Dose Broccoli Sprout vs Low Dose Broccoli Sprout; The null hypothesis is that the urinary sulforaphane levels are equal across treatment arms. Sulforaphane metabolite levels were measured daily for 10 days in each arm; Test type: Equivalence — Statistical significance of the treatment effect (p < 0.01) for the lower doses compared to the high dose as the reference; p < 0.001, Mixed Models Analysis — Using a linear mixed effects model with random intercepts and slope, SF level (in the log scale) was regressed on categorical treatment group (medium dose and low dose; high as the reference) as well as day (continuous variable); Mean Difference (Final Values) = -1.73, 95% CI 2-sided [-1.89 to -1.57], Standard Error of Mean 0.090

2. Secondary Outcome: Modulation of Air Pollutant Excretion in Sequential Overnight 12-Hour Urine Samples
Description: Benzene-mercapturic acid (SPMA) excretion was measured in the sequential overnight 12-hour urine samples collected across the 10-day study period. Data from each individual were summed and averaged to provide a single "per 12-hours" value for each participant.
Time Frame: 10 days
Population: Due to irreversible failure of the mass spectrometer used in this analysis, not all urine samples were evaluated for SPMA levels. Only individuals for whom all 10 samples were collected and analyzed are included in this summary (132/169).
Measure: Geometric Mean (Inter-Quartile Range); unit: nmol SPMA excreted/ 12 hours
Arm/Group | Placebo | Low Dose Broccoli Sprout | Medium Dose Broccoli Sprout | High Dose Broccoli Sprout
Number analyzed (Participants) | 42 | 44 | 26 | 20
nmol SPMA excreted/ 12 hours | 0.67 [0.43 to 0.97] | 0.62 [0.39 to 1.02] | 0.74 [0.62 to 1.18] | 1.09 [0.67 to 1.64]
Statistical Analysis 1: Comparison: Placebo vs Low Dose Broccoli Sprout vs Medium Dose Broccoli Sprout vs High Dose Broccoli Sprout; All broccoli sprout arms were compared with the placebo arm; Test type: Superiority — To summarize first 12-hour SPMA levels over the study course by participant, the SPMA geometric mean (in the log scale) for each individual was calculated and used as the outcome. Treatment arms (placebo, fifth, half and full doses) were independent (categorical) variables in a linear regression model with placebo as the reference; p < 0.05, Regression, Linear; Mean Difference (Final Values) = 63.2, 95% CI 2-sided [10.6 to 140.9] — This Estimation Parameter was based on the comparison between the full dose group and the placebo group

ADVERSE EVENTS:
Time Frame: Daily during the course of the 10-day study and again 1 week after completion of the study
Arm/Group | Placebo | High Dose Broccoli Sprout | Medium Dose Broccoli Sprout | Low Dose Broccoli Sprout
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/25 | 0/35 | 0/55
Other Adverse Events (participants affected / at risk) | 0/55 | 0/25 | 0/35 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No